CLINICAL TRIAL: NCT01900314
Title: Imaging Biomarkers for TMS Treatment of Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Neuronetics (Other)
Responsible Party: Principal Investigator, Stephan Taylor, Professor of Psychiatry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: HUM00053677; 1R21MH098174-01A1 (NIH)
Record Dates: First submitted 2013-07-11; First posted 2013-07-16 (Estimated); Results first posted 2017-04-25 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Depression
Keywords: Major Depression; Major Depressive Disorder; TMS; rTMS
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active rTMS (Active Comparator): 20 active sessions, within a 4 week period, where subjects receive the same repetitive Transcranial Magnetic Stimulation (rTMS) treatment parameters as the FDA-approved device label (10 Hz) to a targeted area of the brain. After these sessions, a second fMRI will be completed then 5 additional tapering treatments of rTMS over a 2 week period.
  Interventions: Device: repetitive Transcranial Magnetic Stimulation (rTMS)
- Sham rTMS (Sham Comparator): 20 sham sessions, within a 4 week period, where subjects receive inactive treatments (0 Hz) of repetitive Transcranial Magnetic Stimulation (rTMS). After 20 sessions and completion of a second fMRI scan, patients in this group will then be unblinded and transitioned to the active arm and will receive a full course (25 sessions) of active rTMS over a 6 week period.
  Interventions: Device: repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: repetitive Transcranial Magnetic Stimulation (rTMS) — 20 active sessions, within a 4 week period, where subjects receive the same repetitive Transcranial Magnetic Stimulation (rTMS) treatment parameters as the sham arm.
  Other Names: TMS; NeuroStar; Sham treatment

SUMMARY:
The purpose of this research is to learn more about how rTMS works to reduce the symptoms of depression. This information can be used to improve the effectiveness of the treatment. The study will use functional magnetic resonance imaging (fMRI) to examine changes in brain function after treatment with rTMS. fMRI is a safe and painless technique that allows investigators to observe the brain "at work." The investigators will use fMRI to see what regions of the brain become active when you perform a concentration task and how that activation is changed after rTMS.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of major depressive disorder
* Male and female subjects, ages 22-65
* Have failed at least 1 antidepressant medication at adequate dose and duration
* On stable antidepressant medication regimen for at least 4 weeks prior to TMS therapy

Exclusion Criteria:

* Diagnosed with a psychotic, bipolar, obsessive-compulsive or post-traumatic stress disorder
* Active substance abuse, including alcohol
* Medical and/or neurological condition that could affect your brain function or risk of seizure, including a stroke, epilepsy, or a closed head injury;
* No presence of an implanted device like a pacemaker/neurostimulator or metal in the head or body;
* Pregnant or trying to get pregnant
* Failed to respond to an adequate course of electroconvulsive therapy (ECT)
* Previous treatment with TMS
* Current depressive episode longer than 5 years

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-09; Primary Completion 2016-01 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan F Taylor, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Taylor SF, Ho SS, Abagis T, Angstadt M, Maixner DF, Welsh RC, Hernandez-Garcia L. Changes in brain connectivity during a sham-controlled, transcranial magnetic stimulation trial for depression. J Affect Disord. 2018 May;232:143-151. doi: 10.1016/j.jad.2018.02.019. Epub 2018 Feb 21. PMID 29494898

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited between October 2013 and October 2015. Subjects exhibited moderate levels of treatment resistance
Pre-assignment Details: 44 patients were screened in person and 40 consented for the study.
Groups:
- Active rTMS: 20 active sessions, within a 4 week period, where subjects receive the same repetitive Transcranial Magnetic Stimulation (rTMS) treatment parameters as the FDA-approved device label (10 Hz) to a targeted area of the brain. After these sessions, a second functional magnetic resonance imaging scan will be completed then 5 additional tapering treatments of rTMS over a 2 week period.
  repetitive Transcranial Magnetic Stimulation (rTMS): 20 active sessions, within a 4 week period, where subjects receive the same repetitive Transcranial Magnetic Stimulation (rTMS) treatment parameters as the sham arm.
- Sham rTMS: 20 sham sessions, within a 4 week period, where subjects receive inactive treatments (0 Hz) of repetitive Transcranial Magnetic Stimulation (rTMS). After 20 sessions and completion of a second functional magnetic resonance imaging scan, patients in this group will then be unblinded and transitioned to the active arm and will receive a full course (25 sessions) of active rTMS over a 6 week period.
  repetitive Transcranial Magnetic Stimulation (rTMS): 20 active sessions, within a 4 week period, where subjects receive the same repetitive Transcranial Magnetic Stimulation (rTMS) treatment parameters as the sham arm.
Period: Overall Study
Arm/Group | Active rTMS | Sham rTMS
Started | 20 | 20
Completed MRI#1 (MRI required BEFORE first treatment) | 17 (2 withdrew consent prior to MRI, 1 had MRI technical failure) | 17 (2 withdrew consent, 1 patient was unable to tolerate MRI)
Completed | 16 (1 patient had MRI, then moved away after 5 TMS treatments) | 16 (1 patient had 4 TMS Tx, but missed too many for protocol requirements,)
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 3 | 3

BASELINE CHARACTERISTICS:
Population: Baseline data for completers only, since this is the group entered into the analysis.
Groups:
- Active rTMS: 20 active sessions
- Sham rTMS: 20 sham sessions
- Total: Total of all reporting groups
Arm/Group | Active rTMS | Sham rTMS | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.9 (10.7) | 44.1 (11.1) | 45.5 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 5 | 6 | 11
MADRS [Mean (Standard Deviation); unit: units on a scale] — MADRS: Montgomery Asberg Depression Rating Scale Range: 0 - 60 0 to 6 - normal/symptom absent 7 to 19 - mild depression 20 to 34 - moderate depression >34 - severe depression
  units on a scale | 25.4 (5.7) | 21.9 (3.1) | 23.5 (5.1)
HRSD-17 [Mean (Standard Deviation); unit: units on a scale] — Depressive symptoms as measured by the 17-item Hamilton Depression Rating Scale (HRSD17) Range: 0-53 Normal: 0-7 Mild: 8 - 13 Moderate 14 - 18 Severe: 19-22 Very severe > 22
  units on a scale | 16 (3.9) | 13.1 (2.3) | 14.2 (4.4)
Global assessment of Function (GAF) [Mean (Standard Deviation); unit: units on a scale] — Range: 0 - 100
  Severely impaired: < 30 moderate impaired: 30-50 mild impaired: 50- 80 No impairment: > 80
  units on a scale | 52.6 (4.7) | 55.6 (4.3) | 54.1 (4.6)
Antidepressant Treatment History Form (ATHF-current) [Mean (Standard Deviation); unit: units on a scale] — ATHF is obtained from interview and review of all treatments, with scores obtained based on the type, duration and length of treatment. This figure represents total number of medications and acceptable augmentation strategies, for the current episode.
  Range: 0 - infinite
  Interpretations: More is worse
  units on a scale | 2.56 (1.75) | 2.94 (1.77) | 2.75 (1.74)

OUTCOME MEASURES:

1. Primary Outcome: Depressive Symptoms at 4 Weeks
Description: MADRS: Montgomery Asberg Depression Rating Scale Range: 0 - 60 0 to 6 - normal/symptom absent 7 to 19 - mild depression 20 to 34 - moderate depression >34 - severe depression
Time Frame: 4 weeks after baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Active rTMS: 20 active sessions of rTMS
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 16 | 16
units on a scale | 15.6 (8.3) | 15.6 (8.3)
Statistical Analysis 1: Comparison: Active rTMS vs Sham rTMS; Repeated measures ANCOVA at 4 weeks with baseline MADRS as co-variate; Test type: Superiority or Other; p = 0.16, ANCOVA

2. Secondary Outcome: Depression Symptoms at 4 Weeks- Secondary
Description: Depressive symptoms as measured by the 17-item Hamilton Depression Rating Scale (HRSD17) Range: 0-53 Normal: 0-7 Mild: 8 - 13 Moderate 14 - 18 Severe: 19-22 Very severe > 22
Time Frame: 4 weeks after baseline
Population: Sample analyzed included all participants who entered the study and received MRI scans at baseline and after 4 weeks of treatment. Repeated measures ANCOVA with screening MADRS score as co-variate
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 16 | 16
units on a scale | 9.1 (4.8) | 10.1 (5.2)
Statistical Analysis 1: Comparison: Active rTMS vs Sham rTMS; Repeated measures ANCOVA with baseline MADRS as co-variate; Test type: Superiority or Other; p = 0.04, ANCOVA

ADVERSE EVENTS:
Time Frame: Adverse events assessed during 4 weeks of double-blinded treatment
Arm/Group | Active rTMS | Sham rTMS
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 4/17 | 5/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active rTMS (N=17) | Sham rTMS (N=17)
Pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Fatigue (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (Nervous system disorders) | 2 (3) | 1 (1)
parathesia (Nervous system disorders) | 2 (3) | 0 (0)
Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
lower extremity swelling (Skin and subcutaneous tissue disorders) | 1 (1) | 0
URI symptoms (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Small size, not powered for group differences. Primary measure was not clinical, but brain changes (primary measures for this report have only focused on clinical changes as neural changes cannot be entered into this reporting format

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less